CLINICAL TRIAL: NCT05650957
Title: PRactice of VENTilation in Patients With ARDS Due to COVID-19 Versus ARDS Due to Other Pulmonary Infections (PRoVENT-COP)
Brief Title: PRactice of VENTilation in Patients With ARDS Due to COVID-19 vs Pneumonia
Acronym: PRoVENT-COP
Status: Completed | Type: Observational
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Collaborators: Carlos III Health Institute (Other Government); University of Sao Paulo (Other); National University of Ireland, Galway, Ireland (Other); Amsterdam UMC (Other)
Responsible Party: Principal Investigator, Prof. Dr. Marcus J. Schultz, Prof. Dr., Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Other Study IDs: AUMC
Record Dates: First submitted 2022-12-13; First posted 2022-12-14 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Acute Respiratory Distress Syndrome; COVID-19; Pneumonia; Mechanical Ventilation Complication
Keywords: Mechanical ventilation; Acute Respiratory Distress Syndrome; Ventilation practice; Pulmonary infection; COVID-19
MeSH Terms: conditions — Respiratory Distress Syndrome; COVID-19; Pneumonia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Non-COVID-19 ARDS: To be included in this analysis the cause for ARDS was a pulmonary infection other than COVID-19 and meeting all aspects of the Berlin definition.
- COVID-19 ARDS: To be included in this analysis the cause for ARDS was COVID-19 and meeting all aspects of the Berlin definition.

SUMMARY:
This study aims to compare epidemiology, management of invasive ventilation and outcomes in critically ill patients with COVID-19 ARDS and ARDS from another pulmonary infection. The investigators will use individual patient data from four recently published large observational COVID-9 studies, including the 'Practice of VENTilation in COVID-19 patients' (PRoVENT-COVID) study, the 'Epidemiology of COVID-19 patients in the ICU' (EPICCoV) study, the 'SATI-COVID-19 - Clinical Characteristics and Outcomes of Patients With COVID-19 on Mechanical Ventilation in Argentina: a Prospective, Multicenter Cohort Study' and the CIBERESUCICOVID - Personalized Risk and Prognosis Factors and Follow-up at One Year of the Patients Hospitalized in the Spanish Intensive Care Units Infected with COVID -19' study. The investigators will use the individual patient data from ARDS patients with another pulmonary infection from the 'LUNG -SAFE - Large Observational Study to UNderstand the Global Impact of Severe Acute Respiratory FailurE' study and the 'ERICC - Epidemiology of Respiratory Insufficiency in Critical Care' study.

DETAILED DESCRIPTION:
Early on in the pandemic, it was frequently proposed that ARDS caused by COVID-19 and ARDS caused by another cause were distinct in a number of ways. COVID-19 related ARDS phenotypes have been suggested, based on differences in respiratory system compliance (Crs) and the severity of the hypoxemia. Other reports have even suggested that lung-protective ventilation strategies for patients with ARDS caused by COVID-19 should differ from those used before the pandemic.

The use of low tidal volumes (VT) and prone positioning, which have been shown to be useful in reducing death in patients with ARDS prior to the pandemic, were also shown to be effective in patients with COVID-19 related ARDS, according to several reports. In the discussion of how to ventilate patients with COVID-19 related ARDS, the disagreement over other ventilatory settings, such as the best positive end-expiratory pressure (PEEP) and the use of recruitment manoeuvres, remains remarkably lively.

To compare epidemiology, management of invasive ventilation and outcomes in critically ill patients with COVID-19 ARDS and ARDS from another pulmonary infection, the investigators will use individual patient data from PRoVENT-COVID, EPICCoV, SATI-COVID-19, CIBERESUCICOVID, LUNG-SAFE and ERICC.

ELIGIBILITY:
Inclusion Criteria:

1. Cause for ARDS is COVID -19 (confirmed with polymerase chain reaction (PCR) and/or presence of typical abnormalities on chest computer tomography (CT) and/or X-ray) or a pulmonary infection from another origen
2. Meeting a Berlin criteria for ARDS
3. Invasive ventilation

Exclusion Criteria:

1. Age < 18 years
2. Any form of non-invasive ventilation

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult critically ill patients receiving invasive ventilation due to ARDS caused by COVID -19 or a pulmonary infection from another origen.
Sampling Method: Non-Probability Sample
Enrollment: 7145 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2024-02-01 (Actual); Study Completion 2024-02-01 (Actual)

PRIMARY OUTCOMES:
Characteristics of invasive ventilation | Day 1
  A combination of key ventilation characteristics, including tidal volume (VT); positive end-expiratory pressure (PEEP); fraction inspired oxygen (FiO2); peak pressure (Ppeak) and plateau pressure (Pplat); respiratory rate (RR); driving pressure (ΔP); respiratory system compliance (CRS) and mechanical power of ventilation (MP).

SECONDARY OUTCOMES:
Ventilator-free days | 28 days
  Liberated of invasive ventilation and alive
Incidence of ICU mortality | 90 days
  Incidence of ICU mortality at day 28 and at day 90
Incidence of in-hospital mortality | 90 days
  Incidence of in-hospital mortality at day 28 and at day 90
ICU length of stay | 90 days
  ICU length of stay at day 28 and at day 90
Hospital length of stay | 90 days
  Hospital length of stay at day 28 and at day 90

CONTACTS AND LOCATIONS:
Overall Officials: David MP van Meenen, PhD, Study Chair — Amsterdam UMC, location AMC
Locations (6):
- Hospital Interzonal General de Agudos'General Jose de San Martin', La Plata, Argentina
- Brazil (2):
  - Hospital Sirio-Libanes, São Paulo
  - Univeristy of São Paulo, São Paulo
- University of Galway, Galway, Ireland
- Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA), Amsterdam, Netherlands
- Carlos III health institute, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Yes
The database will be available after publication of the main publication upon reasonable request after consent of the steering committee. Request must be accompanied by a statistical analysis plan.
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: One year after publication of the main publication
Access Criteria: All requests must be accompanied by a statistical analysis plan

REFERENCES:
- [Derived] van der Ven FLIM, Blok SG, Azevedo LC, Bellani G, Botta M, Estenssoro E, Fan E, Ferreira JC, Laffey JG, Martin-Loeches I, Motos A, Pham T, Penuelas O, Pesenti A, Pisani L, Neto AS, Schultz MJ, Torres A, Tsonas AM, Paulus F, van Meenen DMP; and for the ERICC-; LUNG SAFE-; PRoVENT-COVID-; EPICCoV-; CIBERESUCICOVID-; SATI-COVID-19-investigators. Epidemiology, ventilation management and outcomes of COVID-19 ARDS patients versus patients with ARDS due to pneumonia in the Pre-COVID era. Respir Res. 2024 Aug 17;25(1):312. doi: 10.1186/s12931-024-02910-2. PMID 39153979